CLINICAL TRIAL: NCT02671773
Title: Characterising the Microbiota in Asthma
Acronym: MIA
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 14016
Record Dates: First submitted 2014-09-25; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Asthma
Keywords: Microbiota
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Sputum samples to be retained containing bacterial DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- BTS Step 2 Asthmatic patients: Group of 20 asthmatic patients on British Thoracic Society (BTS) treatment step 2 - regular low dose inhaled corticosteroids (dose of <400 micrograms/day BDP equivalent)
  Interventions: Drug: Inhaled corticosteroid dose/type
- BTS Step 4 Asthmatic patients on treatment with fluticasone: Group of 15 asthmatic patients on British Thoracic Society (BTS) treatment step 4 - high dose inhaled fluticasone (dose of >500 micrograms/day)
  Interventions: Drug: Inhaled corticosteroid dose/type
- BTS Step 4 Asthmatic patients on treatment with budesonide: Group of 15 asthmatic patients on British Thoracic Society (BTS) treatment step 4 - high dose inhaled budesonide (dose of >800 micrograms/day)
  Interventions: Drug: Inhaled corticosteroid dose/type

INTERVENTIONS:
Drug: Inhaled corticosteroid dose/type

SUMMARY:
Previous work has determined that there are significant differences in the communities of bacteria found in the airways of asthmatic patients compared to those found in the airways of healthy people.

It is not yet clear if these bacterial communities are similar in all patients with asthma or if they are different in people with more severe asthma, with different types of asthma or between asthma patients taking different treatment. This is important to know as any differences in the bacteria present between groups may help to explain why people with asthma do not have the same features of disease.

This research aims to determine if there are any differences in the number and type of bacteria found in the airways of asthmatic patients (1) with different severities of asthma and (2) who use different types of inhaled steroid treatment for asthma.

We will do this by detecting the DNA of bacteria present in phlegm samples from these patients. We will also take measurements of the different components of asthma to see if the bacteria are different in people with different types of disease.

As it is not yet clear if the bacteria detected in phlegm samples from one person may differ on different occasions, we will be taking more than one sample from some patients to see how similar this is over time.

DETAILED DESCRIPTION:
The main aim of this project is to determine if microbiota composition is correlated with disease severity (as determined by BTS step). Although initial studies suggest that asthmatics of different severities may have similar microbiota composition, there is no direct evidence to support this assertion. Also, the three main studies in this area so far have all used different sequencing methods, making comparisons difficult.

The relationship between the microbiota composition of different subjects and clinical measures including bronchial hyperreactivity (as measured by methacholine challenge) and pattern of airway inflammation (as measured by sputum differential cell count and exhaled nitric oxide levels) will be investigated further. Comparisons will also be made between samples from asthmatic patients using the inhaled steroid fluticasone and those using budesonide, as there is evidence suggesting that fluticasone leads to an increased risk of pneumonia and non tuberculous mycobacterial disease in certain patient groups. Unpublished data (Astra Zeneca) suggests the excess risk of pneumonia with fluticasone compared to budesonide may be more pronounced after at least 12 months of treatment with inhaled corticosteroid. Microbiota composition of the sputum samples will be evaluated in conjunction with standard microbiological culture of these samples to allow a comparison between these two methods.

In order to assess the reproducibility of the induced sputum method for assessing the lung microbiota, a repeat sputum sample will be taken from a subgroup of 20 patients within 24 hours of the collection of the first sample and compared. A further sample will be taken from this subgroup of patients 2 weeks later to assess the longitudinal stability of the bacterial population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Male or female
* Diagnosis of asthma
* Non-smokers for 10 years and <10 pack year equivalents in total
* BTS Step 2 patients must have been using inhaled steroids at a dose of BDP ≤ 400 mcg/day FP ≤ 200 mcg/day or BUD ≤ 400 mcg/day for at least 1 year
* BTS Step 4 patients must have been using inhaled steroids at a dose of FP ≥ 500 mcg/day or BUD ≥800 mcg/day for at least 1 year as a separate steroid or inhaled steroid/long acting beta agonist combination.

Exclusion Criteria:

* Respiratory infection or antibiotics within last month
* Pregnancy or intent to become pregnant during course of study
* Other respiratory diagnosis
* Post bronchodilator FEV1 of < 60%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult asthmatic patients on Step 2 or Step 4 of the British Thoracic Society Asthma stepwise management protocol for asthma whose details are stored on the Nottingham Respiratory Research Patient Database or who attend respiratory clinics at the Nottingham City Hospital
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Subject sputum microbiota bacterial diversity (richness) (as quantified by mean number of genera) vs subject BTS treatment step | 1 day
Subject sputum microbiota bacterial diversity (as quantified by Simpson's diversity index) vs subject BTS treatment step | 1 day

SECONDARY OUTCOMES:
Subject sputum microbiota bacterial diversity (richness) (as quantified by mean number of genera) vs FEV1 | 1 day
Subject sputum microbiota bacterial diversity (as quantified by Simpson's diversity index) vs FEV1 | 1 day
Subject sputum microbiota bacterial diversity (richness) (as quantified by mean number of genera) vs sputum differential cell count (%eosinophils/%neutrophils) | 1 day
Subject sputum microbiota bacterial diversity (as quantified by Simpson's diversity index) vs sputum differential cell count (%eosinophils/%neutrophils) | 1 day
Subject sputum microbiota bacterial diversity (richness) (as quantified by mean number of genera) vs exhaled nitric oxide level (ppb) | 1 day
Subject sputum microbiota bacterial diversity (as quantified by Simpson's diversity index) vs exhaled nitric oxide level (ppb) | 1 day
Subject sputum microbiota bacterial diversity (richness) (as quantified by mean number of genera) v PC20 (mg/ml) | 1 day
Subject sputum microbiota bacterial diversity (as quantified by Simpson's diversity index) v PC20 (mg/ml) | 1 day
Subject sputum microbiota bacterial diversity (richness) (as quantified by mean number of genera) v Leicester Cough Questionnaire (LCQ) score | 1 day
Subject sputum microbiota bacterial diversity (as quantified by Simpson's diversity index) v Leicester Cough Questionnaire (LCQ) score | 1 day
Subject sputum microbiota bacterial diversity (richness) (as quantified by mean number of genera) v Asthma Control Questionnaire Score | 1 day
Subject sputum microbiota bacterial diversity (as quantified by Simpson's diversity index) v Asthma Control Questionnaire Score | 1 day
Subject sputum microbiota bacterial diversity (richness) (as quantified by mean number of genera) in patients on inhaled fluticasone v same measure in patients on inhaled budesonide | 1 day
Subject sputum microbiota bacterial diversity (as quantified by Simpson's diversity index) in patients on inhaled fluticasone v same measure in patients on inhaled budesonide | 1 day
Subject sputum microbiota bacterial diversity (richness) (as quantified by mean number of genera) v conventional diagnostic microbiological culture (frequency of microbiological cultures reported as positive (%)) | 1 day
Subject sputum microbiota bacterial diversity (as quantified by Simpson's diversity index) v conventional diagnostic microbiological culture (frequency of microbiological cultures reported as positive (%)) | 1 day
Subject sputum microbiota bacterial diversity (richness) (as quantified by mean number of genera) stability over 24 hour period | 2 days
Subject sputum microbiota bacterial diversity (as quantified by Simpson's diversity index) stability over 24 hour period | 2 days
Subject sputum microbiota bacterial diversity (richness) (as quantified by mean number of genera) over 2 week period | 2 weeks
Subject sputum microbiota bacterial diversity (as quantified by Simpson's diversity index) over 2 week period | 2 weeks
Subject sputum bacterial load as per qPCR quantitation (log10 copy numbers/g or similar) vs subject BTS treatment step | 1 day
Subject sputum bacterial load as per qPCR quantitation (log10 copy numbers/g or similar) vs subject BTS treatment step vs FEV1 | 1 day
Subject sputum bacterial load as per qPCR quantitation (log10 copy numbers/g or similar) vs sputum differential cell count (%eosinophils/%neutrophils) | 1 day
Subject sputum bacterial load as per qPCR quantitation (log10 copy numbers/g or similar) vs exhaled nitric oxide level (ppb) | 1 day
Subject sputum bacterial load as per qPCR quantitation (log10 copy numbers/g or similar) vs PC20 (mg/ml) | 1 day
Subject sputum bacterial load as per qPCR quantitation (log10 copy numbers/g or similar) vs Leicester Cough Questionnaire (LCQ) score | 1 day
Subject sputum bacterial load as per qPCR quantitation (log10 copy numbers/g or similar) vs Asthma Control Questionnaire Score | 1 day
Subject sputum bacterial load as per qPCR quantitation (log10 copy numbers/g or similar) in patients on inhaled fluticasone v same measure in patients on inhaled budesonide | 1 day
Subject sputum bacterial load as per qPCR quantitation (log10 copy numbers/g or similar) stability over 24 hour period | 2 days
Subject sputum bacterial load as per qPCR quantitation (log10 copy numbers/g or similar) v conventional diagnostic microbiological culture (frequency of microbiological cultures reported as positive (%)) | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Research Unit, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Derived] Martin MJ, Zain NMM, Hearson G, Rivett DW, Koller G, Wooldridge DJ, Rose G, Gharbia SE, Forbes B, Bruce KD, Harrison TW. The airways microbiome of individuals with asthma treated with high and low doses of inhaled corticosteroids. PLoS One. 2020 Dec 30;15(12):e0244681. doi: 10.1371/journal.pone.0244681. eCollection 2020. PMID 33378384